CLINICAL TRIAL: NCT00479765
Title: A Phase 1 / 2 Dose Escalation Study of Locally-Administered OncoGel™ in Subjects With Recurrent Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor business decision, not based on safety or efficacy data
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR016-CLN-pro002; OGL-109
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Glioblastoma Multiforme; Brain Neoplasms
Keywords: glioblastoma multiforme; recurrent; Phase 1; Phase 2; Phase I; Phase II; brain; cancer; paclitaxel; intracranial; tumor; local; chemotherapy; brain tumor; brain cancer; glioma; OncoGel
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Recurrence; Neoplasms; Glioma | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): OncoGel administered into remaining cavity after surgical resection. Each dose cohort will receive a different volume of OncoGel
  Interventions: Drug: OncoGel (ReGel/Paclitaxel)

INTERVENTIONS:
Drug: OncoGel (ReGel/Paclitaxel) — OncoGel administered into cavity after surgical resection of recurrent glioma. Each subject will receive one dose of OncoGel on the day of surgical resection.

SUMMARY:
OncoGel™ is a new, experimental drug delivery system that allows the slow continuous release of paclitaxel (an approved intravenous anticancer drug), from a gel (ReGel™) over a long period of time. The gel will disappear in 4 to 6 weeks as it releases the paclitaxel.

The purpose of this study is to evaluate the safety and tolerability of OncoGel when placed into the tumor resection cavity in the brain following surgical removal of the tumor. Dose escalation is conducted by gradually increasing the amount of OncoGel placed in the resection cavity in small groups of patients, and watching the patients closely for side effects before moving to the next dose level. The study will also test whether OncoGel helps to prevent or delay the tumor from regrowing.

DETAILED DESCRIPTION:
This study is for patients with recurrent glioblastoma multiforme. Because most recurrences are in the area of the original resection, local delivery of a chemotherapeutic agent may prevent or delay additional recurrences. Paclitaxel has demonstrated activity against 9L glioma tumor lines, but has poor central nervous system penetration after intravenous administration. OncoGel is a new formulation of paclitaxel in a bioerodible gel that can be administered directly to the brain, thereby bypassing the blood-brain barrier.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 to less than 70 years of age
* Radiological evidence on MRI of progressive recurrent malignant glioma that is unilateral, unifocal, supratentorial and of the minimum tumor volume as required per dose level assignment
* Tumor must have a solid contrast enhancing component
* Gross total resection >95% of the recurrence must be planned
* Must have received prior conventional radiation therapy completed >4 weeks before Study Day 1 (ie, day of craniotomy and OncoGel administration)
* Previous cytoreductive surgery or biopsy with pathologic diagnosis of glioblastoma multiforme
* Diagnosis of glioma at the time of debulking surgery for recurrence (by frozen section or squash preparation)
* Life expectancy > 2 months
* KPS greater than or equal to 70
* Using appropriate birth control, if female of child-bearing potential;
* Able and willing to participate in the study by signing the informed consent document

Exclusion Criteria:

* Contrast-enhancing tumor crossing the midline
* Multifocal or non-contiguous tumor resulting in multiple resection cavities
* Evidence of tumor dissemination (ependymal, leptomeningeal)
* Tumors that result in a lobectomy or after resection leave an insufficient residual cavity to receive the expected OncoGel volume
* Expected communication between the ventricle and resection cavity that cannot be repaired
* Involvement of primary sensorimotor cortex in the dominant hemisphere or within 1.5 cm of the optic chiasm, either optic nerve or any other cranial nerve
* Significantly increased intracranial pressure
* Received any type of stereotactic radiosurgery or brachytherapy with the exception of a stereotactic radiosurgery boost as part of the initial radiation therapy
* History of seizures refractory to two or more anticonvulsant medications co-administered at therapeutic levels
* Impaired organ function as evidenced by clinically significant laboratory parameters including but not limited to the following: Hepatic Status: Bilirubin >2.0 mg/dL; Aspartate transaminase (AST) >2.5 times the normal limit; Alanine aminotransferase (ALT) >2.5 times the normal limit. Hematopoietic Status: Absolute neutrophil count (ANC) <1500mm3; Platelet count <100,000/mm3; Hemoglobin < 10 g/dL. Hemostatic: Prothrombin Time (PT) or INR above normal range; Partial Thromboplastin Time (PTT) above normal range; Bleeding Time outside normal range (if performed by hospital). Renal Status: Serum creatinine >2 mg/dL.
* Contraindication to MRI
* Receipt any chemotherapeutic agent within 28 days of Study Day 1 or nitrosourea within 6 weeks of Study Day 1
* Received any intracerebral investigational agent
* Receipt of another investigational drug or device within 28 days of the planned surgery
* Known history of allergy to paclitaxel or any other component of OncoGel
* Pregnant or lactating
* Concurrent life-threatening disease
* Any medical condition or other circumstance that, in the opinion of the Investigator, would make the subject unlikely or unable to successfully complete the study, or would interfere with analysis of study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej S Lesniak, MD, Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - The University of Chicago Brain Tumor Center, Chicago, Illinois
  - The Johns Hopkins University, Baltimore, Maryland
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- OncoGel: OncoGel administered into remaining cavity after surgical resection. Each dose cohort will receive a different volume of OncoGel
  OncoGel (ReGel/Paclitaxel): OncoGel administered into cavity after surgical resection of recurrent glioma. Each subject will receive one dose of OncoGel on the day of surgical resection.
Period: Overall Study
Arm/Group | OncoGel
Started | 4
Completed | 0
Not Completed | 4
Not completed — study terminated | 4

BASELINE CHARACTERISTICS:
Population: Four subjects were dosed with 5% Oncogel prior to study termination.
Groups:
- OncoGel 5mL: OncoGel 5 mL administered into remaining cavity after surgical resection. Each dose cohort will receive a different volume of OncoGel
  OncoGel (ReGel/Paclitaxel): OncoGel administered into cavity after surgical resection of recurrent glioma. Each subject will receive one dose of OncoGel on the day of surgical resection.
Arm/Group | OncoGel 5mL
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 60 [46 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Occurence of Dose-limiting Toxicities (DLTs)
Description: any evidence or sign of a dose-limiting toxicity after administration to determine the maximum tolerated dose (MTD)
Time Frame: 8 weeks
Measure: Number; unit: dose limiting toxicities
Arm/Group | OncoGel 5mL
Number analyzed (Participants) | 4
dose limiting toxicities | 0

ADVERSE EVENTS:
Arm/Group | OncoGel 5mL
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OncoGel 5mL (N=4)
subdural hematoma (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No